CLINICAL TRIAL: NCT03867162
Title: Phase 2 Open-Label Safety and Immunogenicity Study of Tularemia Vaccine, Live, Attenuated (NDBR 101, Lot 4) in Adult Subjects at Risk of Exposure to Tularemia Bacteria
Brief Title: FY15-14: Tularemia Vaccine Protocol (NDBR Lot 4)
Acronym: NDBR
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor terminated this protocol on Dec17, 2021; no subjects have been enrolled
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: US Army Medical Research Institute of Infectious Diseases (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: S-15-23; FY15-14 (Other: USAMRIID); IND 157 (Other: Food and Drug Administration)
Record Dates: First submitted 2019-02-14; First posted 2019-03-07 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Tularemia
MeSH Terms: conditions — Tularemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Live Attenuated Tularemia Vaccine (Experimental): 0.06 mL of Tularemia Vaccine, Live, Attenuated, NDBR 101, Lot 4
  Interventions: Biological: Live Attenuated Tularemia Vaccine

INTERVENTIONS:
Biological: Live Attenuated Tularemia Vaccine — Subjects will be vaccinated with a bifurcated needle; approximately 0.06 mL of the reconstituted vaccine will be placed on the volar surface of the forearm and applied by multiple puncture.

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of the tularemia vaccine, live, attenuated, NDBR 101, Lot 4, and collect data on the incidence of occupational tularemia infection in vaccinated personnel.

DETAILED DESCRIPTION:
This protocol is replacing NCT00787826 (S-09-15; FY07-15)

The study population will consist of USAMRIID and qualified extramural participants who are at risk of exposure to tularemia bacteria. This study will be performed at the USAMRIID SIP Clinic. This open-label study represents a continuation of previous research conducted at USAMRIID.

After the enrollment and approval for participation, each subject will be vaccinated with a bifurcated needle; approximately 0.06 mL of the reconstituted vaccine will be placed on the volar surface of the forearm and applied by multiple puncture. The subject will return for follow-up examination on Days 1 and 2; between Days 5-9, 12-16, and 28-35; and at 6 months (± 14 days) after vaccination for clinical evaluation of AEs and to document responses to the vaccine. Additionally, the subject may be asked to return between Days 56-84 for a repeat titer if indicated and ordered by an investigator on the study. The subject's participation in this study will be considered complete at 6 months ± 14 days after vaccination or revaccination. Following documentation of a positive "take" reaction and a titer showing a ≥ 4-fold increase, routine repeat vaccinations or serosurveillance upon continued exposure to the organism are not included in this protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 to 65 years old at time of consent.
2. If female of childbearing potential, must agree to have a urine pregnancy test on the same day before each vaccine administration. (Exception: documented hysterectomy or ≥ 3 years of menopause.) The results must be negative. Females must agree not to become pregnant for 3 months after receipt of the last study treatment (vaccination).
3. Be considered at risk for exposure to Francisella tularensis (F tularensis) and who have submitted a Request for IND Vaccines for the tularemia vaccine.
4. Sign and date the approved informed consent document and HIPAA Authorization.
5. Have in their charts:

   1. medical history (including concomitant medications) within 60 days of planned first administration of vaccine
   2. physical examination and laboratory tests within 1 year
6. Be medically cleared for participation by an investigator. (Examinations and/or tests may be repeated at the discretion of the principal investigator [PI].)
7. Be willing to return for all follow-up visits.
8. Agree to report any adverse events (AEs) that may or may not be associated with administration of the vaccine for at least 28 days after administration and agree to report all serious adverse events (for example, resulting in hospitalization) for the duration of the subject's participation in the study.
9. Agree to defer blood donation for 1 year after receipt of the vaccine.

Exclusion Criteria:

1. Have been vaccinated against tularemia or had a documented, confirmed tularemia infection.
2. Have received antibiotic therapy within 7 days before vaccination.
3. Have clinically significant abnormal laboratory results (including evidence of hepatitis C, hepatitis B carrier state) or elevated liver function tests (2 times the normal range or at the discretion of the PI). All abnormal laboratory values will be discussed with the research monitor and documented before a subject is enrolled in the trial.
4. Have a personal history of an immunodeficiency, splenectomy or received treatment with an immunosuppressive medication, such as systemically administered glucocorticoids (eg prednisone) within 1 month before planned administration of the vaccine or with other immunosuppressive therapies within 6 months of planned administration of the vaccine. Other immunosuppressive therapies include all cancer chemotherapeutic agents, drugs to prevent transplant rejection, interferons, monoclonal antibodies, protein kinase inhibitors, methotrexate, TNF (tumor necrosis factor) inhibitors, and any other drug determined to be immunosuppressive by the PI. Current administration of topical, inhalational, or intranasal glucocorticoids is not excluded.
5. Have confirmed HIV infection.
6. Have a positive pregnancy test or be a breastfeeding female.
7. Have any known allergies to components of the vaccine:

   1. Live, attenuated Francisella tularensis
   2. Modified casein partial hydrolysate (MCPH) broth
   3. Glucose cysteine hemin agar (GCHA)
   4. Sucrose Gelatin Agar Stabilizer
8. Have administration of blood products (such as blood transfusion, platelet transfusion, immunoglobulin and/or hyperimmune serum), another vaccine or investigational product within 28 days of tularemia vaccination.
9. Have any unresolved AE resulting from a previous immunization.
10. Have an acute or chronic medical condition (such as acute/chronic kidney disease, pulmonary disease, metabolic disease, skin disease) that, in the judgment of the PI, would impact subject safety.

    -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06-09 (Estimated); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
Number of erythematous papule, vesicle and/or eschar with or without underlying induration | 7 days after vaccination
  Incidence of positive "take" reaction (development of an erythematous papule, vesicle, and/or eschar with or without underlying induration )following vaccination for all subjects regardless of compliance
Microagglutination (MA) titer that shows a greater than or equal to 4 fold rise in antibody titer after vaccination | 28-35 days after vaccination
  Seroconversion will be evaluated for subjects who are compliant with the titer schedule

SECONDARY OUTCOMES:
Number of tularemia cases following exposure to F. tularensis in a successfully vaccinated individual | 5 years
  Documented occurrence of tularemia following exposure to F. tularensis in a successfully vaccinated (positive "take" reaction and seroconversion)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin C Pierson, MD, Principal Investigator — USAMRIID
Locations (1):
- Special Immunizations Program, Division of Medicine, USAMRIID, Fort Deterick, Maryland, United States

IPD SHARING:
Plan to Share IPD: No